CLINICAL TRIAL: NCT04091893
Title: The Analgesic Museum: The Development and Effectiveness of Museum-Based Experiences to Reduce Social Isolation and Pain Among Individuals With Chronic Pain
Brief Title: The Development and Effectiveness of Museum-Based Experiences for Individuals With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1415639
Record Dates: First submitted 2019-09-06; First posted 2019-09-17 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Due to covid the in-person RCT was suspended and transitioned to virtual museum programming. Twenty-seven individuals were randomized into the in-person study and 122 individuals were randomized into the virtual study for a total of 149 enrolled individuals.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual care/wait list (Active Comparator)
  Interventions: Behavioral: Usual care/wait list
- Art Rx (Experimental)
  Interventions: Behavioral: Art Rx
- Artful Meditation (Experimental)
  Interventions: Behavioral: Artful Meditation
- Art Rx + Artful Meditation (Experimental)
  Interventions: Behavioral: Art Rx; Behavioral: Artful Meditation

INTERVENTIONS:
Behavioral: Usual care/wait list — Individuals in this group can continue with their usual care (but receive no museum-based intervention)
  Arms: Usual care/wait list
Behavioral: Art Rx — Individuals in this group participate in a specialized tour of an art museum
  Arms: Art Rx; Art Rx + Artful Meditation
Behavioral: Artful Meditation — Individuals in this group participate in a meditation and art appreciation program at an art museum
  Arms: Art Rx + Artful Meditation; Artful Meditation

SUMMARY:
Aim 1: To conduct a formative evaluation of museum-based programming to address loneliness and social isolation.

Aim 2: To develop a consensus-derived Model Museum-Based Program (MMBP) to address loneliness among individuals with chronic pain.

Aim 3: To evaluate the feasibility of museum experiences to reduce loneliness and pain among isolated individuals with chronic pain.

Due to safety concerns related to the covid pandemic in-person museum programming could not continue and virtual versions of the interventions were created. We will publish results on both the in-person and virtual versions of the intervention as well as a pooled analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English speaking
* Chronic pain (6 months or longer)
* Moderate pain or greater (4/10 or greater on a Numerical Rating Scale, range of 0 (no pain) - 10 (worst pain imaginable), in response to the question "Over the past week what was your average pain intensity?")
* Moderately lonely or greater (Score of 4 or greater on 3 item Loneliness scale, range of 3 - 9)

Exclusion Criteria:

* Participated in an Art Rx tour
* Participated in an Artful Meditation program
* Dementia or Alzheimer's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2019-10-12 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Program satisfaction - quality: NRS | Post-intervention (immediately)
  "Please rate your satisfaction with the overall quality of your experience at the museum?"
  NRS - 0 (extremely dissatisfied) - 10 (extremely satisfied)
Primary clinical outcome for preliminary estimate of efficacy - Social disconnection | Post-intervention (immediately)
  Social disconnection scale; 12 items; scored 1 (not at all) - 5 (very much); range 12-60

SECONDARY OUTCOMES:
Change in pain during intervention: 1=Yes/0=No | Post-intervention (immediately)
  Did you experience any pain relief during the museum experience? 1=Yes/0=No
Percent change in pain during intervention | Post-intervention (immediately)
  If "Yes", what percent pain relief did you receive? 0%-100%
Social disconnection | Post-intervention (immediately)
  Social disconnection scale; 12 items; scored 1 (not at all) - 5 (very much); range 12-60
Pain unpleasantness | Post-intervention (immediately)
  Numerical rating scale (NRS) score of 0 "not unpleasant" - 10 "Most unpleasant sensation imaginable ("intolerable")"
Pain unpleasantness | Post-intervention (3-month follow up)
  Numerical rating scale (NRS) score of 0 "not unpleasant" - 10 "Most unpleasant sensation imaginable ("intolerable")"
Pain intensity: Numerical rating scale (NRS) score | Post-intervention (immediately)
  Numerical rating scale (NRS) score of 0 "no pain" - 10 "worst pain imaginable"
Pain intensity: Numerical rating scale (NRS) score | Post-intervention (3-month follow up)
  Numerical rating scale (NRS) score of 0 "no pain" - 10 "worst pain imaginable"
Pain interference | Post-intervention (3-month follow up)
  PEG scale - a 3 item scale to assess average pain intensity [P], interference with enjoyment of life [E], and interference with general activity [G].
  Item 1: What number best describes your pain on the average in the last week?
  Numerical rating scale (NRS) score of 0 "no pain" - 10 "worst pain imaginable"
  Item 2: What number best describes how, during the past week, pain has interfered with your enjoyment of life?
  Numerical rating scale (NRS) score of 0 "does not interfere" - 10 "completely interferes"
  Item 3: What number best describes how, during the past week, pain has interfered with your general activity?
  Numerical rating scale (NRS) score of 0 "does not interfere" - 10 "completely interferes"
Pain Catastrophizing Scale (PCS) | Post-intervention (3-month follow up)
  The PCS is a 13 item scale, with each item rated on a 5-point scale between: 0 (Not at all) and 4 (all the time). The PCS is broken into three subscales including: magnification, rumination, and helplessness. The total range of scores is between 0-52 with higher values reflecting more salient impacts of pain on one's day to day experience.
Chronic Pain Acceptance Questionnaire 8 (CPAQ-8) | Post-intervention (immediately)
  8 items scale designed to measure acceptance of pain.
  Likert scale 0 (never true) - 6 (always true)
Chronic Pain Acceptance Questionnaire 8 (CPAQ-8) | Post-intervention (3-month follow up)
  8 items scale designed to measure acceptance of pain. Likert scale 0 (never true) - 6 (always true)
PHQ 4 | Post-intervention (3-month follow up)
  4 item scale to measure psychological distress (2 items depression; 2 items anxiety) Likert scale 0 (not at all), 1 (several days), 2 (more than half the days) and 3 (nearly every day)
Program satisfaction - recommend: NRS | Post-intervention (immediately)
  How likely would you be to recommend this program to someone with a similar condition? NRS - 0 (extremely likely) - 10 (extremely unlikely)
Affinity for art | Post-intervention (immediately)
  Participants respond to the following prompt: "I like art" Likert scale: 0 (not at all) - 5 (very much)
Affinity for art | Post-intervention (3-month follow up)
  Participants respond to the following prompt: "I like art" Likert scale: 0 (not at all) - 5 (very much)

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Ambulatory Care Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No